CLINICAL TRIAL: NCT00528047
Title: A Phase I, Multi-center, Open-Label, Dose-Escalation, Safety, Pharmacodynamic and Pharmacokinetic Study of PRLX 93936 Administered Intravenously Daily for Five Days Followed by a 23-Day Rest Period in Patients With Advanced Solid Tumors
Brief Title: Safety Study of PRLX 93936 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolexys Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRLX93936-0001
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Cancer
Keywords: Cancer; Solid Tumor; Metastatic; Neoplasm, Malignant
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRLX 93936 (Experimental)
  Interventions: Drug: PRLX 93936

INTERVENTIONS:
Drug: PRLX 93936 — PRLX 93936 will be administered intravenously over one hour daily for 5 days.

SUMMARY:
The purpose of this study is to test the safety of PRLX 93936 and see what kind of effect it has on patients and their cancer. This study will also determine the highest dose of PRLX 93936 that can be given without causing adverse side effects and the dose of PRLX 93936 that should be used in future studies.

DETAILED DESCRIPTION:
This study will assess the safety, pharmacokinetics, and pharmacodynamics of PRLX 93936 administered intravenously over 1 hr daily for 5 days in patients with advanced solid tumors. Patients will be evaluated prior to dosing, during dosing and following dosing, on a 28-day cycle. Tumor response will be evaluated every other cycle.

Three patients will be assigned per dose level until the Maximum Tolerated Dose (MTD) is reached or a a Dose-Limited Toxicity (DLT) is encountered. Sequential cohorts of three patients will be treated with escalating doses until the Maximum Tolerated Dose (MTD) is reached.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors
* Tumor progression after receiving standard/approved chemotherapy and for whom no available treatment provides clinical benefit
* One or more metastatic tumors measurable on a CT scan or MRI per RECIST criteria
* ECOG performance 0-1
* Life expectancy of at least 3 months
* Age >/= 18 years
* A negative pregnancy test (if female of child-bearing potential)
* Acceptable liver function:
* Bilirubin </= 1.5 times the Upper Limit of Normal (ULN)
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase </= 2.5 times ULN (if liver metastases are present, then </= 5 times ULN is allowed)
* Acceptable renal function:
* Serum creatinine within normal limits, OR calculated creatinine clearance >/= 60 mL/min/1.73m2 for patients with creatinine levels above institutional normal
* Acceptable hematologic status:
* Granulocyte count >/= 1500 cells/mm3
* Platelet count >/= 100,000 (plt/mm3)
* Hemoglobin >/= 9.0 g/dL
* Urinalysis: no clinically significant abnormalities
* Acceptable coagulation status:
* PT within normal limits
* aPTT within normal limits
* Completed any chemotherapy, major surgery, or irradiation at least four weeks before enrollment in this study (six weeks for mitomycin-C or nitrosoureas, and two weeks for "targeted" therapies such as kinase inhibitors). Patient must have recovered from all toxicities incurred as a result of previous therapy.
* QT intervals of QTC </= 450 msec for men and </= 470 msec for women (as measured by Hodges equation)
* Left ventricular ejection fraction >/= 50% by 2D Echocardiogram (or > institutional lower limits of normal)

Exclusion Criteria:

* NYHA Class III or IV, cardiac disease, myocardial infarction within the past six months, unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or nursing women
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within four weeks prior to study entry (six weeks for mitomycin-C or nitrosoureas and two weeks for targeted therapies such as kinase inhibitors).
* Unwillingness or inability to comply with protocol procedures
* Known current infection with HIV, hepatitis B or hepatitis C
* Currently receiving any other investigational agent
* Currently receiving medications metabolized by the cytochrome P450 3A4 enzyme pathway
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis. Patients with brain metastases which are well controlled (patients not taking dexamethasone or anti-seizure medication >/= three months after treatment) may be enrolled.
* Any other severe concurrent disease, which in the judgement of the investigator would make the patient inappropriate for the study
* Diagnosis of hypertension
* Previously enrolled in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Clinical laboratory tests | Weekly
Vital signs | Daily during dosing, then weekly during followup
Electrocardiograms (ECGs) | Multiple times during dosing, then weekly during followup
Echocardiograms (ECHO) | Baseline and every other cycle

SECONDARY OUTCOMES:
Tumor assessment | Baseline and every other cycle
Blood sampling for pharmacokinetics | Days 1 and 5 of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, M.D., Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare; Peter J. Rosen, M.D., Principal Investigator — Tower Cancer Research Foundation; Andrew Wagner, M.D., Ph.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Dana Farber Cancer Institute, Boston, Massachusetts